CLINICAL TRIAL: NCT05985655
Title: A Phase 1/2 Open-label Multicenter Study to Assess the Safety, Pharmacokinetics, and Anti-tumor Activity of GTAEXS617 in Patients With Advanced Solid Tumors
Brief Title: Study to Assess GTAEXS617 in Participants With Advanced Solid Tumors
Acronym: ELUCIDATE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Exscientia AI Ltd., a wholly owned subsidiary of Recursion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Exscientia AI Limited (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GTAEXS617-001
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC); Pancreatic Adenocarcinoma; Non-small Cell Lung Cancer (NSCLC); Platinum-resistant High-grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers (HGSOC); Hormone Receptor Positive [HR+] and Human Epidermal Growth Factor Receptor 2 Negative [HER2-] Breast Carcinoma; Triple Negative Breast Cancer (TNBC)
Keywords: Advanced Solid Tumor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Fallopian Tube Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Dose Escalation Monotherapy (Experimental): Participants will receive GTAEXS617 oral tablets in increasing doses.
  Interventions: Drug: GTAEXS617
- Phase 1: Dose Escalation Combination Therapy (Experimental): Participants will receive GTAEXS617 oral tablets in increasing doses in combination with standard of care (SoC) treatment.
  Interventions: Drug: GTAEXS617; Drug: SoC
- Phase 2: Dose Expansion Monotherapy (Experimental): Participants will receive GTAEXS617 oral tablets at Recommended Phase 2 Dose (RP2D).
  Interventions: Drug: GTAEXS617
- Phase 2: Dose Expansion Combination Therapy (Experimental): Participants will receive GTAEXS617 oral tablets at RP2D in combination with SoC treatment.
  Interventions: Drug: GTAEXS617; Drug: SoC

INTERVENTIONS:
Drug: GTAEXS617 — Administered as specified in the treatment arm.
  Other Names: REC-617
Drug: SoC — Participants will receive selected SoC regimen (fulvestrant, paclitaxel + bevacizumab, pegylated liposomal doxorubicin, or capecitabine) administered as specified in the treatment arm.
  Arms: Phase 1: Dose Escalation Combination Therapy; Phase 2: Dose Expansion Combination Therapy

SUMMARY:
The primary purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and anti-tumor activity of GTAEXS617 (REC-617) in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Life expectancy > 3 months.
* One of the following histologically or cytologically confirmed advanced solid tumors: head and neck squamous cell carcinoma (HNSCC), pancreatic adenocarcinoma, non-small cell lung cancer (NSCLC), breast carcinoma (hormone receptor-positive [HR+] and Human Epidermal Growth Receptor 2 negative [HER2-] that has progressed to a prior treatment with Cyclin-Dependent Kinase 4 (CDK4)/ Cyclin-Dependent Kinase 6 [CDK6] inhibitor), or platinum-resistant high-grade epithelial ovarian, primary peritoneal, or fallopian tube cancers (HGSOC), or triple negative breast cancer (TNBC).
* Must have disease that is advanced (ie, surgery or radiotherapy are not considered to be potentially curative), recurrent, or metastatic following SoC treatments.
* Adequate hematological, liver, and renal function.
* Must have tumor lesion(s) or metastases amenable to biopsy, excluding bone metastases.

Key Exclusion Criteria:

* Active and clinically significant (CS) infection.
* Refractory nausea and/or vomiting, chronic gastrointestinal disease, or previous significant bowel resection, with CS sequelae that would preclude adequate absorption of GTAEXS617.
* Symptomatic central nervous system (CNS) malignancy or metastases.
* Concurrent active or previous malignancy.
* Prior organ or allogeneic stem-cell transplantation.
* Moderate or severe cardiovascular disease.
* Received anticancer therapy within 28 days or 5 half-lives (whichever is shorter) before the first dose of the study treatment.
* Received treatment with known strong/moderate inhibitors and/or strong inducers of cytochrome P450 3A isoform subfamily (CYP3A) within 14 days or 5 half-lives before the first dose of study treatment.
* Received treatment with known inhibitors or inducers of P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP) within 14 days or 5 half-lives before the first dose of study treatment.
* Received treatment with known substrates of organic anion transporting peptide or BCRP within 14 days or 5 half-lives before the first dose of study treatment.
* Unresolved or unstable serious toxic side-effects of prior chemotherapy or radiotherapy
* Has had or is scheduled to have major surgery <28 days prior to the first dose of study treatment.

Note: Other protocol Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to 2 years
Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs) | Up to 28 days
Phase 2 : Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 2 years

SECONDARY OUTCOMES:
Phase 1: ORR as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 2 years
Maximum Plasma Concentration (Cmax) of GTAEXS617 | Predose up to 24 hours postdose
Time Maximum Plasma Concentration (Tmax) of GTAEXS617 | Predose up to 24 hours postdose
Area under Plasma Concentration Curve From Time Zero to the Last Quantifiable Concentration (AUC0-inf) of GTAEXS617 | Predose up to 24 hours postdose
Duration of Response (DOR) | Up to 2 years
Progression-Free Survival (PFS) | Up to 2 years
Disease Control Rate (DCR) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Exscientia AI Ltd.
Locations (12):
- United States (3):
  - START Midwest, Grand Rapids, Michigan
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
- Belgium (4):
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Antwerp
  - Clinique Universitaires Saint-Luc, Brussels
  - Institute Jules Bordet, Brussels
  - CHU Sart Tilman, Liège
- United Kingdom (5):
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - UCL Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Newcastle Upon Tyne NHS Foundation Trust, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No